CLINICAL TRIAL: NCT04287049
Title: Early Bactericidal Activity of Standard Drugs Used to Treat Mycobacterium Avium Complex: a Pilot Study
Brief Title: A Study of Standard Drugs for Mycobacterium Avium Complex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); American College of Chest Physicians (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00221119; K23AI159145-01A1 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mycobacterium Avium Complex
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14 Day Azithromycin Monotherapy (Experimental): For the first 14 days of therapy, participants will receive Azithromycin 250mg PO daily as monotherapy. Beyond day 14, all participants will receive guideline-based standard multi-drug therapy for Mycobacterium avium lung disease, as dictated by the physicians treating the participants.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 250 mg PO daily
  Other Names: Zithromax

SUMMARY:
To assess the early bactericidal activity of Azithromycin 250mg by mouth daily over the first 14 days of treatment for Mycobacterium avium complex (MAC) lung disease.

DETAILED DESCRIPTION:
This research is being done to better understand several important aspects of treatment of Mycobacterium avium complex (MAC) lung infections using an early bactericidal activity (EBA) study design. MAC is an environmental bacteria that can cause chronic lung infection. Early bactericidal activity is the amount of bacterial killing that occurs during the first few weeks of antibiotic treatment. By collecting information about the EBA of azithromycin for MAC, the investigators will quantify the efficacy of azithromycin against pulmonary MAC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Isolation of M. avium intracellulare complex from a respiratory specimen in the preceding 6 months
* Fulfill American Thoracic Society (ATS)/Infectious Diseases Society of America (IDSA) criteria for MAC lung disease
* Intention by the treating clinician to treat for MAC lung disease.
* Ability to produce a sputum sample of at least 10mL in a 16 hour period
* Signed informed consent by the subject

Exclusion Criteria:

* Prior treatment for pulmonary MAC within the past 6 months
* Pregnancy
* HIV with a cluster of differentiation 4 (CD4) <350
* History of solid organ or hematologic transplant
* Contraindication to azithromycin
* Has any other condition that, in the opinion of the PI, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Change in Mycobacterium avium colony count in sputum | Baseline and Day 14
  The early bactericidal activity of azithromycin for Mycobacterium avium will be determined as the change in Mycobacterium avium colony count (log10 colony forming unit (CFU) per mL) in sputum between baseline and day 14.
Change in time to positivity of Mycobacterium avium growth in the Mycobacterial Growth Indicator Tube (MGIT) | Baseline and Day 14
  The time (hours) to positivity in MGIT of Mycobacterium avium will be compared between Baseline and Day 14.

SECONDARY OUTCOMES:
Change in Mycobacterium avium colony count in sputum | Baseline and Day 7
  The bactericidal activity of multidrug therapy for Mycobacterium avium will be determined as the change in Mycobacterium avium colony count (log10 CFU per mL) in sputum between baseline and day 7.
Change in Mycobacterium avium colony count in sputum | Day 7 to Day 14
  The bactericidal activity of multidrug therapy for Mycobacterium avium will be determined as the change in Mycobacterium avium colony count (log10 CFU per mL) in sputum between day 7 and day 14.
Change in Mycobacterium avium colony count in sputum | Baseline and 2 Months
  The bactericidal activity of multidrug therapy for Mycobacterium avium will be determined as the change in Mycobacterium avium colony count (log10 CFU per mL) in sputum between baseline and 2 months.
Change in time to positivity of Mycobacterium avium growth in MGIT | Baseline and Day 7
  The time (hours) to positivity in MGIT of Mycobacterium avium will be compared between baseline and day 7.
Change in time to positivity of Mycobacterium avium growth in MGIT | Day 7 and Day 14
  The time (hours) to positivity in MGIT of Mycobacterium avium will be compared between day 7 and day 14.
Change in time to positivity of Mycobacterium avium growth in MGIT | Baseline and 2 Months
  The time (hours) to positivity in MGIT of Mycobacterium avium will be compared between baseline and 2 months.
Estimation of plasma azithromycin area-under-the-curve (AUC) following oral dosing azithromycin | Pre-dose, 2, 4 and 6 hours post-dose on day 15, and 2 and 6 hours post-dose on day 29
  Area-under-the-curve (ug/mL*hr) will be predicted from plasma azithromycin levels using population pharmacokinetic modeling methods.
Estimation of maximum plasma concentration (Cmax) of azithromycin | Pre-dose, 2, 4 and 6 hours post-dose on day 15
  Peak concentration (Cmax) will be predicted from plasma drug concentration in ug/mL following oral dosing of azithromycin.
Estimation of maximum plasma concentration (Cmax) of azithromycin | 2 and 6 hours post-dose on day 29
  Peak concentration (Cmax) will be predicted from plasma drug concentration in ug/mL following oral dosing of azithromycin.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Ignatius, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Ryu YJ, Koh WJ, Daley CL. Diagnosis and Treatment of Nontuberculous Mycobacterial Lung Disease: Clinicians' Perspectives. Tuberc Respir Dis (Seoul). 2016 Apr;79(2):74-84. doi: 10.4046/trd.2016.79.2.74. Epub 2016 Mar 31. PMID 27066084
- [Background] Griffith DE, Brown BA, Cegielski P, Murphy DT, Wallace RJ Jr. Early results (at 6 months) with intermittent clarithromycin-including regimens for lung disease due to Mycobacterium avium complex. Clin Infect Dis. 2000 Feb;30(2):288-92. doi: 10.1086/313644. PMID 10671330
- [Background] Koh WJ, Moon SM, Kim SY, Woo MA, Kim S, Jhun BW, Park HY, Jeon K, Huh HJ, Ki CS, Lee NY, Chung MJ, Lee KS, Shin SJ, Daley CL, Kim H, Kwon OJ. Outcomes of Mycobacterium avium complex lung disease based on clinical phenotype. Eur Respir J. 2017 Sep 27;50(3):1602503. doi: 10.1183/13993003.02503-2016. Print 2017 Sep. PMID 28954780
- [Background] Asakura T, Nakagawa T, Suzuki S, Namkoong H, Morimoto K, Ishii M, Kurashima A, Betsuyaku T, Ogawa K, Hasegawa N; Nontuberculous Mycobacteriosis Japan Research Consortium (NTM-JRC). Efficacy and safety of intermittent maintenance therapy after successful treatment of Mycobacterium avium complex lung disease. J Infect Chemother. 2019 Mar;25(3):218-221. doi: 10.1016/j.jiac.2018.07.021. Epub 2018 Aug 29. PMID 30172726
- [Background] Jindani A, Aber VR, Edwards EA, Mitchison DA. The early bactericidal activity of drugs in patients with pulmonary tuberculosis. Am Rev Respir Dis. 1980 Jun;121(6):939-49. doi: 10.1164/arrd.1980.121.6.939. No abstract available. PMID 6774638
- [Background] Diacon AH, Dawson R, von Groote-Bidlingmaier F, Symons G, Venter A, Donald PR, van Niekerk C, Everitt D, Winter H, Becker P, Mendel CM, Spigelman MK. 14-day bactericidal activity of PA-824, bedaquiline, pyrazinamide, and moxifloxacin combinations: a randomised trial. Lancet. 2012 Sep 15;380(9846):986-93. doi: 10.1016/S0140-6736(12)61080-0. Epub 2012 Jul 23. PMID 22828481
- [Background] Donald PR, Diacon AH. The early bactericidal activity of anti-tuberculosis drugs: a literature review. Tuberculosis (Edinb). 2008 Aug;88 Suppl 1:S75-83. doi: 10.1016/S1472-9792(08)70038-6. PMID 18762155
- [Background] Slaats MH, Hoefsloot W, Magis-Escurra C, Boeree MJ, Wattenberg M, Kuipers S, van Ingen J. Regimens for nontuberculous mycobacterial lung disease lack early bactericidal activity. Eur Respir J. 2016 Mar;47(3):1000-2. doi: 10.1183/13993003.00925-2015. Epub 2015 Dec 2. No abstract available. PMID 26647433
- [Background] Wallace RJ Jr, Brown BA, Griffith DE, Girard WM, Murphy DT, Onyi GO, Steingrube VA, Mazurek GH. Initial clarithromycin monotherapy for Mycobacterium avium-intracellulare complex lung disease. Am J Respir Crit Care Med. 1994 May;149(5):1335-41. doi: 10.1164/ajrccm.149.5.8173775.